CLINICAL TRIAL: NCT01646476
Title: Comparison of Efficacy of Covered Versus Uncovered Self-expandable Metallic Stents for Treatment of Malignant Gastric Outlet Obstruction: a Prospective, Randomized Study
Brief Title: Covered Versus Uncovered Self-expandable Metallic Stents for Malignant Gastric Outlet Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-01-075
Record Dates: First submitted 2012-07-09; First posted 2012-07-20 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Gastric Outlet Obstruction Due to Gastric Adenocarcinoma
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Covered stent (Bona stent, pyloric/duodenal covered) (Active Comparator): WAVE covered self-expandable metallic stent (BONASTENT, Standard Sci Tech, Ltd., Seoul, Korea)
  Interventions: Device: Covered stent (Bona stent pyloric/duodenal covered) insertion
- Uncovered stent (Bona stent, pyloric/duodenal) (Active Comparator): uncovered self-expandable metallic stent (BONASTENT, Standard Sci Tech, Ltd., Seoul, Korea)
  Interventions: Device: Uncovered stent (Bona stent, pyloric/duodenal) insertion

INTERVENTIONS:
Device: Covered stent (Bona stent pyloric/duodenal covered) insertion — self-expandable metallic stent placement was performed with a therapeutic endoscope (working channel ≥ 3.7 mm) using a through-the-scope method. All patients underwent procedures under conscious sedation with midazolam and pethidine. The length of the stricture was assessed either endoscopically or fluoroscopically; the length of the stent had to exceed that of the stricture by at least 3 cm. After the required stent length was determined, the stent was advanced through the endoscope over a guidewire until it passed across the distal end of the stricture. Then, the stent was deployed under continuous fluoroscopic control. For the Wave covered stent group, the stent was repositioned after deployment using the lasso under fluoroscopic guidance (if necessary), aligning the central portion of the stricture with the central portion of the stent which had reduced radial force and indentation. Stent positioning was confirmed endoscopically and fluoroscopically.
  Arms: Covered stent (Bona stent, pyloric/duodenal covered)
Device: Uncovered stent (Bona stent, pyloric/duodenal) insertion — Self-expandable metallic stent placement was performed with a therapeutic endoscope (working channel ≥ 3.7 mm) using a through-the-scope method. All patients underwent procedures under conscious sedation with midazolam and pethidine. The length of the stricture was assessed either endoscopically or fluoroscopically; the length of the stent had to exceed that of the stricture by at least 3 cm. After the required stent length was determined, the stent was advanced through the endoscope over a guidewire until it passed across the distal end of the stricture. Then, the stent was deployed under continuous fluoroscopic control. For the Wave covered stent group, the stent was repositioned after deployment using the lasso under fluoroscopic guidance (if necessary), aligning the central portion of the stricture with the central portion of the stent which had reduced radial force and indentation. Stent positioning was confirmed endoscopically and fluoroscopically.
  Arms: Uncovered stent (Bona stent, pyloric/duodenal)

SUMMARY:
Malignant gastric outlet obstruction can result from gastric adenocarcinoma, leading to intractable vomiting, nausea, and poor oral food intake. Although self-expandable metallic stent (SEMS) insertion has excellent technical and clinical success rates for relieving gastric outlet obstruction symptoms, the uncovered SEMS is susceptible to re-stenosis because of tumor ingrowth through openings between the stent wire filaments. Therefore, the most common reason for stent failure in uncovered stents is tumor ingrowth.

The covered SEMS has a membrane that prevents ingrowth through the mesh wall and consequently shows lower rate of re-stenosis than uncovered SEMS. However, covered SEMS has a higher risk of stent migration compared to uncovered SEMS. Recent prospective, randomized study showed that there was no significant difference between uncovered and covered SEMS in terms of stent patency rate as well as technical and clinical success rates.

Recently the investigators developed new covered SEMS for gastric outlet obstruction. This new covered SEMS has features that may contribute to reducing migration rate: 1) partially covered design; 2)less radial force in central portion of stent; 3) presence of lasso which enable position of stent to be adjusted after deployment; 4)presence of protrusion in both sides of stent. This prospective, randomized study aimed to compare the effectiveness and side effects of newly developed covered SEMS with those of uncovered SEMS in patients with malignant gastric outlet obstruction from gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* age: 20-80
* patients with gastric outlet obstruction due to gastric adenocarinoma
* patients with inoperable gastric adenocarcinoma due to distant metastasis or severe comorbidity
* Gastric outlet obstruction score: 0-2
* Symptoms consistent with gastric outlet obstruction such as nausea or vomiting
* Findings consistent with gastric outlet obstruction in upper endoscopy or abdominal computed tomography

Exclusion Criteria:

* Previous history of stent insertion or endoscopic dilation for gastric outlet obstruction
* previous history of bypass surgery for gastric outlet obstruction
* Multiple level of bowel obstruction confirmed in radiographic studies such as small bowel series or abdominal computed tomography
* Borrmann type IV advanced gastric cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stent patency | 8 weeks after stent insertion

SECONDARY OUTCOMES:
Stent patency | 16 weeks after stent insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea